CLINICAL TRIAL: NCT05840445
Title: Efficacy of Prabotulinum Toxin-A and Onabotulinum Toxin-A for the Treatment of Expression Lines in the Upper Third of the Face.
Brief Title: Efficacy of Prabotulinum and Onabotulinum Toxin-A for Facial Wrinkles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-026-2020
Record Dates: First submitted 2023-04-11; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Face; Skin Fold; Rejuvenation
Keywords: Botulinum Toxin; Onabotulinum; Prabotulinum; Upper Third Facial Wrinkles; Botulinum Toxin Comparison; Aesthetic
MeSH Terms: conditions — Facies | interventions — onabotulinum toxin A; Botulinum Toxins, Type A; prabotulinumtoxin A

STUDY DESIGN:
Intervention Model Description: Simple randomization was performed in two groups: the Onabotulinum group and the Prabotulinum group. Each group would receive an intramuscular application of onabotulinum toxin-A and prabotulinum toxin-A in the upper facial third, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Onabotulinum Group (Placebo Comparator): This group received an intramuscular application of onabotulinum toxin-A in the upper facial third.
  Interventions: Drug: Onabotulinum toxin A
- Prabotulinum Group (Active Comparator): This group received an intramuscular application of prabotulinum toxin-A in the upper facial third.
  Interventions: Drug: Prabotulinumtoxin A

INTERVENTIONS:
Drug: Onabotulinum toxin A — Intramuscular application of onabotulinum toxin-A in the upper facial third.
  Other Names: Botox
  Arms: Onabotulinum Group
Drug: Prabotulinumtoxin A — Intramuscular application of prabotulinum toxin-A in the upper facial third.
  Other Names: Nabota
  Arms: Prabotulinum Group

SUMMARY:
The appearance of facial wrinkles, lines, or folds is a natural phenomenon during aging. Different scales help classify wrinkles objectively, such as the Facial Wrinkle Scale. Others help classify patients' subjective perspectives, like the Face-Q questionnaire. The application of Botulinum Toxin is the most performed non-surgical aesthetic procedure in the world to treat facial expression lines. The present study aims to compare the efficacy of onabotulinum toxin-A (BOTOX®) and prabotulinum toxin-A (NABOTA®) to treat expression lines in the upper third of the face, based on objective and subjective follow-up, using the FWS scale and FACE-Q questionnaire, respectively.

DETAILED DESCRIPTION:
This is an experimental, comparative, longitudinal, open-label, prospective study at the Instituto de Oftalmología Fundación Conde de Valenciana I.A.P, Mexico City, Mexico.

The investigators used a proportion formula to calculate the sample size, with an alpha value of 0.05, and a precision of 3%. The difference in the effect between the two toxins is 20%, considering a 20% loss, with a total of 18 patients. A nonprobabilistic sampling of consecutive cases was performed. Once patients were selected and included in the study, they were randomly assigned to a group.

After inclusion, simple randomization was performed in the Onabotulinum and Prabotulinum groups. Each group received intramuscular administration of onabotulinum toxin-A and prabotulinum toxin-A in the upper facial third.

The investigators used descriptive statistics to analyze the demographic variables and employed the Mann-Whitney U test to assess differences in the quantitative and ordinal outcome variables between the groups before and at the end of the study. Additionally, the investigators employed the chi-square test to compare the intergroup results before and at the end of the study for nominal variables. To compare intragroup results over time, the investigators conducted a repeated measures ANOVA test for continuous variables, Friedman test for ordinal variables, and Cochran's Q test for nominal variables. We used SPSS Version 20 (Chicago, IL, USA) for analysis and considered a value of p<0.05 as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 25 and 40 years of age
* Diagnosis of expression lines in the upper facial third of any degree
* Wished to improve their aesthetic appearance

Exclusion Criteria:

* Known allergy to milk protein or albumin
* Pregnancy and lactation
* Cardiovascular or neuromuscular disease
* Recent history of infections in the facial region
* Concomitant intake of aminoglycosides or cyclosporine A

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Change in subjective evaluation of botulinum toxin between groups | Pre treatment
  Evaluation using Face-Q questionnaire on each visit, answered by the patient. Questionnaire-based Likert scale with a min value of 1 and maximum value of 4, qualifying patient's satisfaction with their facial appearance.
Change in subjective evaluation of botulinum toxin between groups | On day 7
  Evaluation using Face-Q questionnaire on each visit, answered by the patient. Questionnaire-based Likert scale with a min value of 1 and maximum value of 4, qualifying patient's satisfaction with their facial appearance.
Change in subjective evaluation of botulinum toxin between groups | On day 30
  Evaluation using Face-Q questionnaire on each visit, answered by the patient. Questionnaire-based Likert scale with a min value of 1 and maximum value of 4, qualifying patient's satisfaction with their facial appearance.
Change in subjective evaluation of botulinum toxin between groups | On day 120
  Evaluation using Face-Q questionnaire on each visit, answered by the patient. Questionnaire-based Likert scale with a min value of 1 and maximum value of 4, qualifying patient's satisfaction with their facial appearance.
Change in objective evaluation of botulinum toxin between groups | Pretreatment
  Evaluation using Facial Wrinkle Scale on each visit, made by the main author. It is an objective scale with four points, minimum score 0, none; 1, mild; 2, moderate; and maximum score 3, severe.
Change in objective evaluation of botulinum toxin between groups | On day 7
  Evaluation using Facial Wrinkle Scale on each visit, made by the main author. It is an objective scale with four points, minimum score 0, none; 1, mild; 2, moderate; and maximum score 3, severe.
Change in objective evaluation of botulinum toxin between groups | On day 30
  Evaluation using Facial Wrinkle Scale on each visit, made by the main author. It is an objective scale with four points, minimum score 0, none; 1, mild; 2, moderate; and maximum score 3, severe.
Change in objective evaluation of botulinum toxin between groups | On day 120
  Evaluation using Facial Wrinkle Scale on each visit, made by the main author. It is an objective scale with four points, minimum score 0, none; 1, mild; 2, moderate; and maximum score 3, severe.

SECONDARY OUTCOMES:
Duration of activity | On day 30
  Time of efficacy for muscle blockage on maximun expression
Duration of activity | On day 120
  Time of efficacy for muscle blockage on maximun expression
Onset of action | On day 7
  Time required from application to muscle blockage on maximum expression

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Garfias, PhD, Study Chair — Instituto de Oftalmología Conde de Valenciana I. A. P
Locations (2):
- Mexico (2):
  - Institute of Ophthalmology, Conde de Valenciana Foundation, Mexico City, Mexico City
  - Instituto de Oftalmología, Mexico City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hadi H, Wilkinson CM. Categorizing facial creases: A review. J Cosmet Dermatol. 2017 Jun;16(2):180-185. doi: 10.1111/jocd.12305. Epub 2017 Feb 1. PMID 28145033
- [Background] Yaar M, Gilchrest BA. Photoageing: mechanism, prevention and therapy. Br J Dermatol. 2007 Nov;157(5):874-87. doi: 10.1111/j.1365-2133.2007.08108.x. Epub 2007 Aug 17. PMID 17711532
- [Background] Kohl E, Steinbauer J, Landthaler M, Szeimies RM. Skin ageing. J Eur Acad Dermatol Venereol. 2011 Aug;25(8):873-84. doi: 10.1111/j.1468-3083.2010.03963.x. Epub 2011 Jan 24. PMID 21261751
- [Background] Conkling N, Bishawi M, Phillips BT, Bui DT, Khan SU, Dagum AB. Subjective rating of cosmetic treatment with botulinum toxin type A: do existing measures demonstrate interobserver validity? Ann Plast Surg. 2012 Oct;69(4):350-5. doi: 10.1097/SAP.0b013e31824a43e0. PMID 22964674
- [Background] Sundaram H, Signorini M, Liew S, Trindade de Almeida AR, Wu Y, Vieira Braz A, Fagien S, Goodman GJ, Monheit G, Raspaldo H; Global Aesthetics Consensus Group. Global Aesthetics Consensus: Botulinum Toxin Type A--Evidence-Based Review, Emerging Concepts, and Consensus Recommendations for Aesthetic Use, Including Updates on Complications. Plast Reconstr Surg. 2016 Mar;137(3):518e-529e. doi: 10.1097/01.prs.0000475758.63709.23. PMID 26910696
- [Background] Satriyasa BK. Botulinum toxin (Botox) A for reducing the appearance of facial wrinkles: a literature review of clinical use and pharmacological aspect. Clin Cosmet Investig Dermatol. 2019 Apr 10;12:223-228. doi: 10.2147/CCID.S202919. eCollection 2019. PMID 31114283
- [Background] Huang W, Foster JA, Rogachefsky AS. Pharmacology of botulinum toxin. J Am Acad Dermatol. 2000 Aug;43(2 Pt 1):249-59. doi: 10.1067/mjd.2000.105567. PMID 10906647
- [Background] Klein AW. Contraindications and complications with the use of botulinum toxin. Clin Dermatol. 2004 Jan-Feb;22(1):66-75. doi: 10.1016/j.clindermatol.2003.12.026. PMID 15158548
- [Result] Nam HS, Park YG, Paik NJ, Oh BM, Chun MH, Yang HE, Kim DH, Yi Y, Seo HG, Kim KD, Chang MC, Ryu JH, Lee SU. Efficacy and safety of NABOTA in post-stroke upper limb spasticity: a phase 3 multicenter, double-blinded, randomized controlled trial. J Neurol Sci. 2015 Oct 15;357(1-2):192-7. doi: 10.1016/j.jns.2015.07.028. Epub 2015 Jul 21. PMID 26233808
- [Result] Won CH, Kim HK, Kim BJ, Kang H, Hong JP, Lee SY, Kim CS. Comparative trial of a novel botulinum neurotoxin type A versus onabotulinumtoxinA in the treatment of glabellar lines: a multicenter, randomized, double-blind, active-controlled study. Int J Dermatol. 2015 Feb;54(2):227-34. doi: 10.1111/ijd.12627. Epub 2014 Oct 14. PMID 25311357
- [Result] Cheon HI, Jung N, Won CH, Kim BJ, Lee YW. Efficacy and Safety of Prabotulinumtoxin A and Onabotulinumtoxin A for Crow's Feet: A Phase 3, Multicenter, Randomized, Double-Blind, Split-Face Study. Dermatol Surg. 2019 Dec;45(12):1610-1619. doi: 10.1097/DSS.0000000000001920. PMID 30893169